CLINICAL TRIAL: NCT01128894
Title: A Randomized, Open-Label, Parallel-Group, Multicenter Study to Determine the Efficacy and Safety of Albiglutide as Compared With Liraglutide in Subjects With Type 2 Diabetes Mellitus
Brief Title: A Study to Determine the Efficacy and Safety of Albiglutide as Compared With Liraglutide.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 114179
Record Dates: First submitted 2010-04-29; First posted 2010-05-24 (Estimated); Results first posted 2014-05-20 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-01

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: GSK716155; liraglutide; albiglutide; open-label
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — rGLP-1 protein; Liraglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- albiglutide (Experimental): weekly albiglutide subcutaneous injection
  Interventions: Biological: albiglutide
- liraglutide (Active Comparator): liraglutide daily subcutaneous injection, starting at 0.6mg, then up-titrating to 1.2mg then 1.8mg in accordance with prescribing information.
  Interventions: Drug: liraglutide

INTERVENTIONS:
Biological: albiglutide — albiglutide weekly subcutaneous injection
  Arms: albiglutide
Drug: liraglutide — liraglutide daily subcutaneous injection, starting at 0.6mg, then up-titrating to 1.2mg then 1.8mg in accordance with prescribing information.
  Arms: liraglutide

SUMMARY:
This open-label study examines the efficacy and safety of albiglutide as compared with liraglutide in subjects with type 2 diabetes.

DETAILED DESCRIPTION:
This randomized, open-label, multicenter, 2 parallel-group study evaluates the efficacy and safety of a weekly subcutaneously injected dose of albiglutide as compared with liraglutide. Subjects with a historical diagnosis of type 2 diabetes mellitus and whose glycemia is inadequately controlled on their current regimen of metformin, thiazolidinedione, sulfonylurea, or any combination of these oral antidiabetics will be recruited into the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 2 diabetes mellitus and experiencing inadequate glycemic control on their current regimen of metformin, TZD, SU, or any combination of these oral antidiabetic medications
* BMI >/=20kg/m2 and </=45 kg/m2
* Fasting C-peptide >/=0.8 ng/mL (>/=0.26 nmol/L)
* HbA1c between 7.0% and 10.0%, inclusive
* Female subjects of childbearing potential must be practicing adequate contraception.

Exclusion Criteria:

* History of cancer
* History of treated diabetic gastroparesis
* Current biliary disease or history of pancreatitis
* History of significant GI surgery
* Recent clinically significant cardiovascular and/or cerebrovascular disease
* Hypertension
* History of human immunodeficiency virus infection
* History of or current liver disease or acute symptomatic infection with hepatitis B or hepatitis C
* History of alcohol or substance abuse
* Female subject is pregnant, lactating, or <6 weeks postpartum
* Known allergy to any GLP 1 analogue, liraglutide, other study medications' excipients, excipients of albiglutide, or Baker's yeast
* History of type 1 diabetes mellitus
* Contraindications (as per the prescribing information) for the use of either background or potential randomized study medications (e.g., liraglutide)
* Receipt of any investigational drug or liraglutide within the 30 days or 5 half lives, whichever is longer, before Screening or a history of receipt of an investigational antidiabetic drug within the 3 months before randomization or receipt of albiglutide in previous studies
* History or family history of thyroid disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 841 (Actual)
Dates: Start 2010-05; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (150):
- United States (111):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Chandler, Arizona
  - GSK Investigational Site, Gilbert, Arizona
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Searcy, Arkansas
  - GSK Investigational Site, Chula Vista, California
  - GSK Investigational Site, Escondido, California
  - GSK Investigational Site, Fresno, California
  - GSK Investigational Site, Huntington Beach, California
  - GSK Investigational Site, Indio, California
  - GSK Investigational Site, Irvine, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Mission Viejo, California
  - GSK Investigational Site, Orange, California
  - GSK Investigational Site, Palm Desert, California
  - GSK Investigational Site, Riverside, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Satna Monica, California
  - GSK Investigational Site, Spring Valley, California
  - GSK Investigational Site, Tarzana, California
  - GSK Investigational Site, Tustin, California
  - GSK Investigational Site, Walnut Creek, California
  - GSK Investigational Site, West Hills, California
  - GSK Investigational Site, Clearwater, Florida
  - GSK Investigational Site, Cocoa, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, North Miami, Florida
  - GSK Investigational Site, Ocala, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Pembroke Pines, Florida
  - GSK Investigational Site, St. Petersburg, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Winter Park, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Blue Ridge, Georgia
  - GSK Investigational Site, Roswell, Georgia
  - GSK Investigational Site, Stone Mountain, Georgia
  - GSK Investigational Site, Honolulu, Hawaii
  - GSK Investigational Site, Idaho Falls, Idaho
  - GSK Investigational Site, La Grange, Illinois
  - GSK Investigational Site, Evansville, Indiana
  - GSK Investigational Site, Valparaiso, Indiana
  - GSK Investigational Site, Council Bluffs, Iowa
  - GSK Investigational Site, Dubuque, Iowa
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, Paducah, Kentucky
  - GSK Investigational Site, Covington, Louisiana
  - GSK Investigational Site, Shreveport, Louisiana
  - GSK Investigational Site, Haverhill, Massachusetts
  - GSK Investigational Site, Bloomfield Hills, Michigan
  - GSK Investigational Site, Dearborn, Michigan
  - GSK Investigational Site, Detroit, Michigan
  - GSK Investigational Site, Kalamazoo, Michigan
  - GSK Investigational Site, Saint Clair Shores, Michigan
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Picayune, Mississippi
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Lincoln, Nebraska
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Elizabeth, New Jersey
  - GSK Investigational Site, Haddon Heights, New Jersey
  - GSK Investigational Site, North Massapequa, New York
  - GSK Investigational Site, Staten Island, New York
  - GSK Investigational Site, Burlington, North Carolina
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Greensboro, North Carolina
  - GSK Investigational Site, Lenoir, North Carolina
  - GSK Investigational Site, Morehead City, North Carolina
  - GSK Investigational Site, Shelby, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Canal Fulton, Ohio
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Dayton, Ohio
  - GSK Investigational Site, Gallipolis, Ohio
  - GSK Investigational Site, Kettering, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Downington, Pennsylvania
  - GSK Investigational Site, Greer, South Carolina
  - GSK Investigational Site, Murrells Inlet, South Carolina
  - GSK Investigational Site, Simpsonville, South Carolina
  - GSK Investigational Site, Bristol, Tennessee
  - GSK Investigational Site, Clarksville, Tennessee
  - GSK Investigational Site, Memphis, Tennessee
  - GSK Investigational Site, Tullahoma, Tennessee
  - GSK Investigational Site, Arlington, Texas
  - GSK Investigational Site, Corpus Christi, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Hurst, Texas
  - GSK Investigational Site, Katy, Texas
  - GSK Investigational Site, Midland, Texas
  - GSK Investigational Site, North Richland Hills, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Schertz, Texas
  - GSK Investigational Site, Sugarland, Texas
  - GSK Investigational Site, Bountiful, Utah
  - GSK Investigational Site, Draper, Utah
  - GSK Investigational Site, West Jordan, Utah
  - GSK Investigational Site, South Burlington, Vermont
  - GSK Investigational Site, Burke, Virginia
  - GSK Investigational Site, Manassas, Virginia
  - GSK Investigational Site, Richmond, Virginia
  - GSK Investigational Site, Salem, Virginia
  - GSK Investigational Site, Spokane, Washington
  - GSK Investigational Site, Tacoma, Washington
- Australia (9):
  - GSK Investigational Site, Garran, Australian Capital Territory
  - GSK Investigational Site, Camperdown, New South Wales
  - GSK Investigational Site, St Leonards, New South Wales
  - GSK Investigational Site, Herston, Queensland
  - GSK Investigational Site, Box Hill, Victoria
  - GSK Investigational Site, Geelong, Victoria
  - GSK Investigational Site, Heidelberg, Victoria
  - GSK Investigational Site, Ringwood East, Victoria
  - GSK Investigational Site, Fremantle, Western Australia
- Israel (4):
  - GSK Investigational Site, Beersheba
  - GSK Investigational Site, Haifa
  - GSK Investigational Site, Kfar Saba
  - GSK Investigational Site, Nahariya
- Peru (6):
  - GSK Investigational Site, Ica, Ica
  - GSK Investigational Site, Lima, Lima Province
  - GSK Investigational Site, Huacho, Lima region
  - GSK Investigational Site, Callao, Lima
  - GSK Investigational Site, Piura, Piura
  - GSK Investigational Site, Lima
- Philippines (6):
  - GSK Investigational Site, Cebu City
  - GSK Investigational Site, Iloilo City
  - GSK Investigational Site, Makati City
  - GSK Investigational Site, Marikina City
  - GSK Investigational Site, Pasay
  - GSK Investigational Site, Pasig
- South Korea (3):
  - GSK Investigational Site, Goyang
  - GSK Investigational Site, Seongnam-si
  - GSK Investigational Site, Seoul
- Spain (6):
  - GSK Investigational Site, A Coruña
  - GSK Investigational Site, Alicante
  - GSK Investigational Site, Majadahonda (Madrid)
  - GSK Investigational Site, Modulo H
  - GSK Investigational Site, Sabadell
  - GSK Investigational Site, Torrevieja (Alicante)
- United Kingdom (5):
  - GSK Investigational Site, London, London
  - GSK Investigational Site, Birmingham
  - GSK Investigational Site, Hertfordshire
  - GSK Investigational Site, Livingston
  - GSK Investigational Site, Swansea

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Pratley RE, Nauck MA, Barnett AH, Feinglos MN, Ovalle F, Harman-Boehm I, Ye J, Scott R, Johnson S, Stewart M, Rosenstock J; HARMONY 7 study group. Once-weekly albiglutide versus once-daily liraglutide in patients with type 2 diabetes inadequately controlled on oral drugs (HARMONY 7): a randomised, open-label, multicentre, non-inferiority phase 3 study. Lancet Diabetes Endocrinol. 2014 Apr;2(4):289-297. doi: 10.1016/S2213-8587(13)70214-6. Epub 2014 Feb 6. PMID 24703047
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 114179 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 114179 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 114179 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 114179 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 114179 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 114179 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 114179 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Eligible participants entered into 2 weeks of Prescreening and Screening; 4 weeks of Run-in/stabilization; a 32-week Treatment Period for evaluation of efficacy and safety and 8 weeks of post treatment Follow-up. A total of 1764 participants were screened, 841 were randomized and 812 received at least one dose of study treatment.
Groups:
- Albiglutide 50 mg: Participants received albiglutide 30 milligrams (mg) once weekly subcutaneously (SC) from Baseline until Week 6 with up-titration to 50 mg weekly at Week 6.
- Liraglutide 1.8 mg: Participants received liraglutide 0.6 mg once daily (OD) SC from Baseline until Week 1. From Week 1 to Week 2 the dose was increased to 1.2 mg. At Week 2, the dose was increased to 1.8 mg.
Period: Overall Study
Arm/Group | Albiglutide 50 mg | Liraglutide 1.8 mg
Started | 404 | 408
Completed | 346 | 340
Not Completed | 58 | 68
Not completed — Adverse Event | 31 | 41
Not completed — Protocol Violation | 2 | 1
Not completed — Noncompliance | 4 | 5
Not completed — Lost to Follow-up | 8 | 8
Not completed — Withdrawal by Subject | 10 | 12
Not completed — Physician Decision | 2 | 1
Not completed — Conflicting HbA1c Results at Screening | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Albiglutide 50 mg | Liraglutide 1.8 mg | Total
Number analyzed (Participants) | 404 | 408 | 812
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.4 (10.11) | 55.8 (9.95) | 55.6 (10.03)
Gender [Count of Participants; unit: Participants]
  Female | 213 | 190 | 403
  Male | 191 | 218 | 409
Race/Ethnicity, Customized [Number; unit: Participants]
  African American/African Heritage | 47 | 29 | 76
  American Indian or Alaskan Native | 30 | 37 | 67
  Asian - Central/South Asian Heritage | 3 | 9 | 12
  Asian - East Asian Heritage | 26 | 18 | 44
  Asian - Japanese Heritage | 0 | 3 | 3
  Asian - South East Asian Heritage | 17 | 19 | 36
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  White - Arabic/North African Heritage | 5 | 6 | 11
  White - White/Caucasian/European Heritage | 276 | 285 | 561

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Glycosylated Hemoglobin (HbA1c) at Week 32
Description: HbA1c is a form of hemoglobin that is measured primarily to identify the average plasma glucose concentration over a 2- to 3-month period. The Baseline HbA1c value is defined as the last non-missing value before the start of treatment. Change from Baseline in HbA1c was calculated as the value at Week 32 minus the value at Baseline. The analysis was performed using an Analysis of Covariance (ANCOVA) model with treatment group, region, history of prior myocardial infarction (yes versus no), and age category (<65 years versus ≥65 years) as factors and Baseline HbA1c as a continuous covariate. The last observation carried forward (LOCF) method was used to impute missing data, in which the last non-missing post-Baseline on-treatment measurement was used to impute the missing measurement. If a participant had missing observation(s) immediately after Baseline, the Baseline observation was not carried forward and was left as missing.
Time Frame: Baseline and Week 32
Population: Intent-to-Treat (ITT) Population: all participants who received at least one dose of study medication and who had at least one post-Baseline assessment of the primary endpoint, HbA1c. Only those participants available at the indicated time point were assessed.
Measure: Least Squares Mean (Standard Error); unit: Percentage of HbA1c in the blood
Arm/Group | Albiglutide 50 mg | Liraglutide 1.8 mg
Number analyzed (Participants) | 398 | 402
Percentage of HbA1c in the blood | -0.78 (0.047) | -0.99 (0.046)
Statistical Analysis 1: Comparison: Albiglutide 50 mg vs Liraglutide 1.8 mg; Test type: Non-Inferiority or Equivalence — The p-value was from a 1-sided t test testing whether or not the difference of least square means (albiglutide - liraglutide) was less than or equal to the prespecified noninferiority margin of 0.3%; p = 0.0846, ANCOVA; Mean Difference (Final Values) = 0.21, 95% CI 2-sided [0.08 to 0.34]

2. Secondary Outcome: Mean Change From Baseline in HbA1c at Weeks 4, 6, 12, 18 and 26
Description: HbA1c is a form of hemoglobin that is measured primarily to identify the average plasma glucose concentration over a 2- to 3-month period. The Baseline HbA1c value is defined as the last non-missing value before the start of treatment. Change from Baseline was calculated as the post-Baseline value minus the Baseline value. The LOCF method was used to impute missing data, in which the last non-missing post-Baseline on-treatment measurement was used to impute the missing measurement. If a participant had missing observation(s) immediately after Baseline, the Baseline observation was not carried forward and was left as missing. Participants were considered in the treatment week if they had received at least one dose in that treatment week.
Time Frame: Baseline, Weeks 4, 6, 12, 18 and 26
Population: ITT Population. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles). Different participants may have been analyzed at different time points, so the overall number of participants analyzed reflects everyone in the ITT Population.
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c in the blood
Arm/Group | Albiglutide 50 mg | Liraglutide 1.8 mg
Number analyzed (Participants) | 402 | 403
Percentage of HbA1c in the blood
  Week 4, n=387, 392 | -0.52 (0.481) | -0.73 (0.447)
  Week 6, n=398, 401 | -0.66 (0.566) | -0.94 (0.569)
  Week 12, n=398, 402 | -0.88 (0.824) | -1.18 (0.798)
  Week 18, n=398, 402 | -0.87 (0.921) | -1.13 (0.904)
  Week 26, n=398, 402 | -0.79 (0.968) | -1.00 (0.969)

3. Secondary Outcome: Mean Change From Baseline in Fasting Plasma Glucose (FPG) at Week 32
Description: The FPG test measures blood sugar levels after the participant has not eaten (fasted) for 12 to 14 hours. The Baseline FPG value is the last non-missing value before the start of treatment. Change from Baseline was calculated as the post-Baseline value minus the value at Baseline. The analysis was performed using an Analysis of Covariance (ANCOVA) model with treatment group, region, Baseline HbA1c category, history of prior myocardial infarction (yes versus no), and age category (<65 years versus ≥65 years) as factors and Baseline FPG as a continuous covariate. The LOCF method was used to impute missing data, in which the last non-missing post-Baseline on-treatment measurement was used to impute the missing measurement. If a participant had missing observation(s) immediately after Baseline, the Baseline observation was not carried forward and was left as missing. Participants were considered in the treatment week if they had received at least one dose in that treatment week.
Time Frame: Baseline and Week 32
Population: ITT Population. Only those participants available at the indicated time point were assessed.
Measure: Least Squares Mean (Standard Error); unit: Millimoles per liter (mmol/L)
Arm/Group | Albiglutide 50 mg | Liraglutide 1.8 mg
Number analyzed (Participants) | 400 | 402
Millimoles per liter (mmol/L) | -1.22 (0.115) | -1.68 (0.115)

4. Secondary Outcome: Mean Change From Baseline in Fasting Plasma Glucose (FPG) at Weeks 1, 2, 3, 4, 6, 12, 18 and 26
Description: The FPG test measures blood sugar levels after the participant has not eaten (fasted) for 12 to 14 hours. The Baseline FPG value is the last non-missing value before the start of treatment. Change from Baseline was calculated as the post-Baseline value minus the value at Baseline. The LOCF method was used to impute missing data, in which the last non-missing post-Baseline on-treatment measurement was used to impute the missing measurement. If a participant had missing observation(s) immediately after Baseline, the Baseline observation was not carried forward and was left as missing. Participants were considered in the treatment week if they had received at least one dose in that treatment week.
Time Frame: Baseline, Weeks 1, 2, 3, 4, 6, 12, 18 and 26
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Millimoles per liter (mmol/L)
Arm/Group | Albiglutide 50 mg | Liraglutide 1.8 mg
Number analyzed (Participants) | 402 | 403
Millimoles per liter (mmol/L)
  Week 1, n=386, 381 | -0.98 (1.939) | -1.62 (2.116)
  Week 2, n= 399, 398 | -1.33 (2.194) | -2.25 (2.296)
  Week 3, n= 400, 402 | -1.61 (2.067) | -2.43 (2.470)
  Week 4, n= 400, 402 | -1.52 (2.148) | -2.45 (2.381)
  Week 6, n= 400, 402 | -1.25 (2.317) | -2.11 (2.451)
  Week 12, n= 400, 402 | -1.73 (2.526) | -2.10 (2.590)
  Week 18, n= 400, 402 | -1.44 (2.362) | -1.74 (2.704)
  Week 26, n= 400, 402 | -1.14 (2.694) | -1.64 (2.717)

5. Secondary Outcome: Number of Participants Who Achieved HbA1c Response Level of <6.5% and <7.0% at Week 32
Description: Number of participants who achieved HbA1c response levels of <6.5% and <7.0% at Week 32 were assessed. The last observation carried forward (LOCF) method was used to impute missing data, in which the last non-missing post-Baseline on-treatment measurement was used to impute the missing measurement. If a participant had missing observation(s) immediately after Baseline, the Baseline observation was not carried forward and was left as missing.
Time Frame: Week 32
Population: ITT Population. Only those participants available at the indicated time point were assessed.
Measure: Number; unit: Participants
Arm/Group | Albiglutide 50 mg | Liraglutide 1.8 mg
Number analyzed (Participants) | 398 | 402
Participants
  HbA1c <6.5% | 78 | 113
  HbA1c <7.0% | 168 | 208

6. Secondary Outcome: Time to Hyperglycemia Rescue at Week 32
Description: Participants who experienced persistent hyperglycemia (high blood glucose) could have qualified for hyperglycemia rescue. The conditions for hyperglycemia rescue were as follows: fasting plasma glucose (FPG) >=280 milligram/decilitre (mg/dL) >= Week 2 and < Week 4, FPG >=250 mg/dL >= Week 4 and <Week 12, HbA1c ≥8.5% and ≤0.5% reduction from Baseline- >= Week 12 and <Week 26, or HbA1c ≥8.5% >= Week 26. Time to hyperglycemia rescue is defined as the time between the date of the first dose of study medication and the date of hyperglycemia rescue plus one day, or the time between the date of the first dose of study medication and the date of the last visit during the active treatment period plus one day for participants not requiring rescue. This time was divided by 7 to express the result in weeks. All times extending beyond Week 32 relevant to hyperglycemia rescue were censored at Week 32.
Time Frame: Week 32
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Albiglutide 50 mg | Liraglutide 1.8 mg
Number analyzed (Participants) | 402 | 403
Weeks | NA [NA to NA] — There were too few events of hyperglycemia rescue (<50% of participants with events) to calculate the median and confidence interval. | NA [NA to NA] — There were too few events of hyperglycemia rescue (<50% of participants with events) to calculate the median and confidence interval.

7. Secondary Outcome: Mean Change From Baseline in Body Weight at Week 32
Description: The Baseline value is the last non-missing value before the start of treatment. Change from Baseline was calculated as the value at Week 32 minus the value at Baseline. The analysis was performed using an Analysis of Covariance (ANCOVA) model with treatment group, region, Baseline HbA1c category, history of prior myocardial infarction (yes versus no), and age category (<65 years versus ≥65 years) as factors and Baseline weight as a continuous covariate. The LOCF method was used to impute missing data, in which the last non-missing post-Baseline on-treatment measurement was used to impute the missing measurement. If a participant had missing observation(s) immediately after Baseline, the Baseline observation was not carried forward and was left as missing. Weight values obtained after hyperglycemia rescue were treated as missing and replaced with pre-rescue values.
Time Frame: Baseline and Week 32
Population: ITT Population. Only those participants available at the indicated time point were assessed.
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Albiglutide 50 mg | Liraglutide 1.8 mg
Number analyzed (Participants) | 400 | 402
Kilograms | -0.62 (3.118) | -2.21 (4.147)

ADVERSE EVENTS:
Time Frame: On-treatment serious adverse events (SAEs) and non-serious adverse events (AEs), defined as those events occurring while participants were on treatment up until 56 days after the last dose (up to Week 40), are reported.
Description: SAEs and AEs were collected in members of the Safety Population, comprised of all participants randomized to treatment, who received at least one dose of the study medication.
Arm/Group | Albiglutide 50 mg | Liraglutide 1.8 mg
Serious Adverse Events (participants affected / at risk) | 20/404 | 23/408
Other Adverse Events (participants affected / at risk) | 266/404 | 289/408
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Albiglutide 50 mg (N=404) | Liraglutide 1.8 mg (N=408)
Atrial fibrillation (Cardiac disorders) | 2 | 2
Myocardial infarction (Cardiac disorders) | 1 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 0
Atrial flutter (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1
Coronary artery occlusion (Cardiac disorders) | 0 | 1
Gastroenteritis (Infections and infestations) | 2 | 0
Cellulitis (Infections and infestations) | 0 | 1
Encephalitis herpes (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 1 | 0
Pneumonia viral (Infections and infestations) | 1 | 0
Tracheobronchitis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 1 | 0
Chest pain (General disorders) | 1 | 2
Non-cardiac chest pain (General disorders) | 1 | 1
Pyrexia (General disorders) | 1 | 0
Sudden death (General disorders) | 0 | 1
Convulsion (Nervous system disorders) | 0 | 2
Transient ischaemic attack (Nervous system disorders) | 2 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Ileus (General disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Burns first degree (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Renal colic (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0
Arteriosclerosis (Vascular disorders) | 1 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 1
Retinal detachment (Eye disorders) | 0 | 1
Hepatitis (Hepatobiliary disorders) | 1 | 0
Blood amylase increased (Investigations) | 0 | 1
Lipase increased (Investigations) | 0 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Albiglutide 50 mg (N=404) | Liraglutide 1.8 mg (N=408)
Diarrhoea (Gastrointestinal disorders) | 60 | 55
Nausea (Gastrointestinal disorders) | 40 | 119
Vomiting (Gastrointestinal disorders) | 20 | 38
Constipation (Gastrointestinal disorders) | 17 | 25
Dyspepsia (Gastrointestinal disorders) | 17 | 25
Abdominal pain upper (Gastrointestinal disorders) | 11 | 10
Abdominal distension (Gastrointestinal disorders) | 11 | 8
Abdominal pain (Gastrointestinal disorders) | 10 | 11
Flatulence (Gastrointestinal disorders) | 10 | 9
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 9 | 14
Upper respiratory tract infection (Infections and infestations) | 42 | 45
Urinary tract infection (Infections and infestations) | 25 | 23
Nasopharyngitis (Infections and infestations) | 24 | 28
Sinusitis (Infections and infestations) | 12 | 7
Bronchitis (Infections and infestations) | 11 | 9
Influenza (Infections and infestations) | 7 | 13
Gastroenteritis (Infections and infestations) | 7 | 11
Hypoglycaemia (Metabolism and nutrition disorders) | 66 | 83
Decreased appetite (Metabolism and nutrition disorders) | 12 | 28
Injection site reaction (General disorders) | 28 | 5
Fatigue (General disorders) | 13 | 10
Injection site haematoma (General disorders) | 7 | 9
Oedema peripheral (General disorders) | 4 | 10
Headache (Nervous system disorders) | 22 | 22
Dizziness (Nervous system disorders) | 10 | 21
Arthralgia (Musculoskeletal and connective tissue disorders) | 16 | 12
Back pain (Musculoskeletal and connective tissue disorders) | 15 | 19
Lipase increased (Investigations) | 22 | 28
Hypertension (Vascular disorders) | 13 | 15
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 12
Anaemia (Blood and lymphatic system disorders) | 5 | 10
Contusion (Injury, poisoning and procedural complications) | 5 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.